CLINICAL TRIAL: NCT01304251
Title: Effects of Short-term Fasting on Tolerance to Adjuvant Chemotherapy in Breast Cancer Patients
Brief Title: Effects of Short-term Fasting on Tolerance to Chemotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, Hanno Pijl, Prof. dr. H. Pijl, Leiden University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: P10.247
Record Dates: First submitted 2011-02-24; First posted 2011-02-25 (Estimated); Last update posted 2016-01-12 (Estimated); Status verified 2016-01

CONDITIONS: Breast Cancer
Keywords: short-term fasting; adjuvant chemotherapy; toxicity; side-effects
MeSH Terms: conditions — Breast Neoplasms; Intermittent Fasting | interventions — Diet, Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Short-term fasting (Active Comparator): short term fasting (i.e. 24 hours before and 24 hours after administration of chemotherapy) in 20 breast cancer patients
  Interventions: Other: Short-term fasting
- Healthy nutrition (Placebo Comparator): 20 breast cancer patients eat according to the current guidelines for healthy nutrition as from 24 hours before until 24 hours after the beginning of administration of chemotherapy.
  Interventions: Other: Healthy nutrition

INTERVENTIONS:
Other: Short-term fasting — Short-term fasting, i.e. 24 hours before and 24 hours after administration of chemotherapy
  Arms: Short-term fasting
Other: Healthy nutrition — Eating according to the current guidelines for healthy nutrition as from 24 hours before until 24 hours after the beginning of administration of chemotherapy. Dietary instructions will be given by a dietician and actual food intake will be recorded in a journal.
  Arms: Healthy nutrition

SUMMARY:
The purpose of this study is to determine the effect of short-term fasting on tolerance to adjuvant chemotherapy in breast cancer patients

DETAILED DESCRIPTION:
Evidence from experimental animals provides strong support for the concept that caloric restriction (CR) increases resistance to multiple forms of stress. CR decreases plasma levels of growth factors, e.g. insulin-like growth factor-I (IGF-I), thereby diverting energy from growth to maintenance. Accordingly, the currently available information suggests that short-term fasting protects normal cells against the perils of (high dose) chemotherapy. In contrast, cancer cells are not (or less) protected as a result of their self-sufficiency in growth signals. This phenomenon is termed Differential Stress Resistance (DSR). DSR reduces the severity of side-effects caused by the toxicity of chemotherapy, without interfering with its effect on reduction of tumour volume or tumour markers. A recent report, sketching a case series of 10 cancer patients, suggests that short term fasting protects against the side effects of chemotherapy in humans. Indeed, the majority of patients preferred fasting over feeding in preparation of their therapy. This study aims to further evaluate the impact of fasting on tolerance to chemotherapy in humans.

ELIGIBILITY:
Inclusion Criteria:

* Female breast cancer patients, receiving adjuvant TAC-chemotherapy
* Age ≥ 18 years old
* WHO performance status 0-2
* Adequate bone marrow function: white blood cells (WBCs) ≥ 3.0 x 109/l, neutrophils ≥ 1.5 x 109/l, platelets ≥ 100 x 109/l
* Adequate liver function: bilirubin ≤ 1.5 x upper limit of normal (UNL) range, ALAT and/or ASAT ≤ 2.5 x UNL, Alkaline Phosphatase ≤5 x UNL
* Adequate renal function: the calculated creatinine clearance should be ≥ 50 mL/min
* Survival expectation > 3 months
* Patients must be accessible for treatment and follow-up
* Written informed consent according to the local Ethics Committee requirements

Exclusion Criteria:

* Serious other diseases such as recent myocardial infarction, clinical signs of cardiac failure or clinically significant arrhythmias
* Diabetes Mellitus
* body mass index (BMI) < 19 kg/m2
* Pregnancy or lactating
* Medical or psychological condition which in the opinion of the investigator would not permit the patient to complete the study or sign meaningful informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2011-03; Primary Completion 2013-04 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
chemotherapy-induced neutropenia | approximately 126 days
  Neutrophil count after 6 cycles of chemotherapy (6x 21 days)

SECONDARY OUTCOMES:
chemotherapy-induced DNA damage in leukocytes | 21 days
  chemotherapy-induced DNA damage in leukocytes will be determined after each cycle of chemotherapy (i.e. every 21 days)
perceived side effects of chemotherapy | 21 days
  To determine the effect of short-term fasting on perceived side effects after each cycle of chemotherapy (i.e. every 21 days)
effect of short-term fasting on the body's inflammatory response to chemotherapy | 21 days
  To determine the effect of short-term fasting on the body's inflammatory response to chemotherapy, inflammation parameters will be measured after each cycle of chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Hanno Pijl, MD PhD, Principal Investigator — Leiden University Medical Center
Locations (1):
- Leiden University Medical Center, Leiden, Netherlands

REFERENCES:
- [Result] Safdie FM, Dorff T, Quinn D, Fontana L, Wei M, Lee C, Cohen P, Longo VD. Fasting and cancer treatment in humans: A case series report. Aging (Albany NY). 2009 Dec 31;1(12):988-1007. doi: 10.18632/aging.100114. PMID 20157582
- [Derived] de Groot S, Vreeswijk MP, Welters MJ, Gravesteijn G, Boei JJ, Jochems A, Houtsma D, Putter H, van der Hoeven JJ, Nortier JW, Pijl H, Kroep JR. The effects of short-term fasting on tolerance to (neo) adjuvant chemotherapy in HER2-negative breast cancer patients: a randomized pilot study. BMC Cancer. 2015 Oct 5;15:652. doi: 10.1186/s12885-015-1663-5. PMID 26438237